CLINICAL TRIAL: NCT06693089
Title: Metacognitive Interpersonal Therapy Across Transdiagnostic Eating Disorders Including Underweight: Study Protocol for a Single-arm Pilot Study
Brief Title: Metacognitive Interpersonal Therapy Across Transdiagnostic Eating Disorders, Including Underweight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GLORIA FIORAVANTI (Other)
Collaborators: Simone Cheli (Unknown); Angus MacBeth (Unknown); Francesca Travagnin (Unknown); Martina Nicolis (Unknown); Valentina Nicolosi (Unknown); Raffaele Popolo (Unknown); Giancarlo Dimaggio (Unknown)
Responsible Party: Sponsor-Investigator, GLORIA FIORAVANTI, Gloria Fioravanti, Centro Trattamento Integrato: Disturbi Alimentari e Obesita
Organization: Centro Trattamento Integrato: Disturbi Alimentari e Obesita (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HD7ABEBGC6@ADA91162
Record Dates: First submitted 2024-11-07; First posted 2024-11-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorders; Maladaptive Personality Trait; Personality Disorder; Personality Trait; Emotion Regulation; Social Interaction; Perfectionism; Self Esteem; Cognitive Dysfunction; Dysfunctional Behavior Psychology
Keywords: Mental Disorders; Cognition Disorders; Neurocognitive Disorders; Behavioral Symptoms; Feeding and Eating Disorders; Personality Disorders; Cognitive Dysfunction; Problem Behavior
MeSH Terms: conditions — Feeding and Eating Disorders; Personality Disorders; Emotional Regulation; Cognitive Dysfunction; Problem Behavior; Mental Disorders; Cognition Disorders; Neurocognitive Disorders; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: The study is a single arm study to evaluate MIT-ED effectiveness on a larger sample of adults with transdiagnostic ED presentations which include underweight participants. They will receive up to 40 individual sessions of MIT-ED. The study is run in an private outpatient clinic specialized in eating disorder treatment. Therapies will be delivered both in person or through videoconferencing. Three therapists will be involved in the trial, all trained in MIT.
Masking Description: Treatment-seeking participants will first receive an assessment screening visit. Once evaluated for inclusion/exclusion criteria, and informed written consent has been obtained, baseline measures about primary and secondary outcomes will be completed. Participants will then be proposed for inclusion in the study.
  Recruitment will stop once 64 participants have met inclusion criteria and have accepted to participate to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: MIT-ED (Experimental): Participants will receive 1 or 2 preliminary sessions focused on typical elements of Cognitive Behavioral Therapy for Eating Disorders, including psychoeducational training on eating behaviors, an introduction to tools such as monitoring forms, weight charts, and assessments of eating behaviors like physical exercise, body checking, and episodes of binging, purging, and starvation. Before treatment starts, patients meet with a dietitian to develop a nutritional plan that normalizes calorie intake, which will be reviewed throughout treatment. After these sessions, participants will receive up to 40 weekly individual sessions.
  Given the inclusion of underweight patients, the protocol developed by Fioravanti and colleagues (2023) required adaptations, such as considering the effects of malnutrition on cognitive and organic functioning and extending psychotherapy for up to 40 sessions.
  Interventions: Other: MIT-ED

INTERVENTIONS:
Other: MIT-ED — The aim is to develop healthier strategies for managing negative thoughts and feelings linked to Eating Disorder (ED) and engage patients in social interactions that fulfill their relational needs. Participants will learn that perfectionism and the need for control in ED are coping strategies shaped by interpersonal patterns with significant others, where low self-esteem and emotional dysregulation play key roles. Metacognitive Intepersonal Therapy (MIT) aims to improve individuals' ability to understand their own emotions and thoughts, recognizing maladaptive, rigid, and biased schemas about self and others. This awareness helps them form a richer understanding of others' minds and use this knowledge to respond more adaptively to social challenges. MIT also helps individuals reflect on how these schemas trigger ED behaviors and develop better coping strategies for interpersonal stressors.

SUMMARY:
The goal of this clinical trial is to assess if Metacognitive Interpersonal Therapy for Eating Disorders (MIT-ED) is effective for treating various forms of Eating Disorders (ED) and reducing dropout rates. The trial will also evaluate its feasibility and outcomes in a patient group including also underweight participants. The main questions it aims to answer are:

* Does MIT-ED improve eating disorder symptoms and reduce overall maintenance factors, as alexithymia, emotional dysregulation, maladaptive perfectionism, and self-esteem?
* Is MIT-ED effective in reducing the severity of personality disorders and associated global psychiatric symptoms?
* What are the dropout rates and adherence levels for patients receiving MIT-ED?

Participants will:

* Undergo an initial screening to confirm eligibility, including a comprehensive clinical interview and assessments based on inclusion and exclusion criteria for the study.
* Receive up to 40 individual sessions of MIT-ED, each lasting 50-60 minutes, over a period of approximately 10-12 months.
* Attend regular assessment focusing on eating disorder symptoms (Eating Disorder Examination Questionnaire, EDE-Q 6.0, and ED Interview, EDE), emotional dysregulation (Difficulties in Emotion Regulation Scale, DERS), alexithymia (Toronto Alexithymia Scale-20, TAS-20), and self-esteem (Rosenberg Self-Esteem Scale, RSES). Assessment will be conducted at baseline (before starting MIT-ED sessions), after 20 MIT-ED sessions (approximately after 5 months), post-treatment (approximately after 10 months), and at 3 months follow-up. A longer 12-months follow-up is planned.

Researchers will evaluate the effectiveness of MIT-ED based on treatment adherence, symptom improvement, and the reduction of maintenance mechanisms associated with Eating Disorders. Positive results could support the design of a larger, controlled Randomized Clinical Trial (RCT).

DETAILED DESCRIPTION:
This is a single arm study. The hypotheses are that Metacognitive Interpersonal Therapy for Eating Disorders (MIT-ED) will be able to keep drop-out lower than possible, estimated <20%; promote remission in the primary Eating Disorder (ED) measure; achieve weight gain in underweight participants.

Recruitment will stop once 64 participants have met inclusion criteria and have accepted to participate to the study. The study will recruit adults aged 18 and over, diagnosed with an ED within the past six months, from the Centro di Trattamento Integrato - Disturbi Alimentari e Obesità (CTI-Disturbi Alimentari e Obesità) in Verona and Genova. Underweight individuals will be included to evaluate MIT-ED's broader applicability.

Participants will receive up to 40 individual sessions of MIT-ED, delivered either in-person or via videoconferencing by 3 trained therapists. Therapists will receive 2 hours supervision every two weeks with 2 of Metacognitive Interpersonal Therapy designers. Therapy sessions will be randomly audio-recorded for process analysis Assessments will occur at baseline, after 20 MIT-ED sessions (approximately after 5 months), post-treatment (approximately after 10 months), and at 3 months follow-up, where publications of the results are scheduled. A longer term 12-months follow-up is planned. A research assistant will handle psychometric test administration and coordination with the clinical team.

This study will provide preliminary evidence on the feasibility and effectiveness of MIT-ED in a broader ED population, including underweight patients. The results will inform the design of a larger controlled trials to further validate MIT-ED efficacy with the hope it results as a new treatment option for patients with transdiagnostic ED.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients (from age 18 years)
* Having an Eating Disorder for which they required treatment
* BMI between 17.5 and 40
* Provision of informed consent

Exclusion Criteria:

* Receiving ongoing psychiatric, other psychotherapeutic treatment
* Coexisting psychiatric disorders precludeing eating disorder-focused treatment or that requires specialized treatment: bipolar I, psychosis, alcohol or substance abuse, suicidality. PTSD is an exclusion criteria as long as its symptoms as prominent so to require a specialized empirically supported treatment
* Intellectual disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q 6.0; Fairburn & Beglin, 1994) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  A self report measure assessing eating disorders over the past 4 weeks, providing a measure of the range of severity of eating disorder features. The questionnaire consists of 28 items with responses ranging from 0 to 6 (where 6 indicates higher gravity of the disorder).
Eating Disorder Examination Interview (EDE, Fairburn, Cooper & O'Connor; 2014). | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  An interview based on the Eating Disorder Examination Questionnaire-6 questionnaire, which provides information about the main behavioural characteristics of eating disorders. Questions concern the frequency in which the patient engages in behaviors indicative of an eating disorder over a 28-day period. The test is scored on a 7-point scale from 0-6. With a zero score indicating not having engaged in the questioned behavior.

SECONDARY OUTCOMES:
Binge Eating Scale (BES; Gormally et al., 1992) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  A self-report questionnaire of the behavioral, cognitive and emotional features of objective binge eating (OBE). The total score ranges from 0 to 46, with higher scores correlating with more frequent and severe binge eating behaviors.
Body Mass Index (BMI) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  As an additional measure of the recovery from eating disorder (BMI <18.5). Body Mass Index is a measure of weight relative to height.
Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Disorders (SCID-5; Michael B. First, Janet B.W. Williams) | At baseline and after 20 sessions of therapy (approximately after 5 months)
  For assessing and defining Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Model for Personality Disorders. The scoring system for the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Disorders (SCID-5) varies depending on the specific disorder being assessed, but generally a minimum score indicates that the criteria for a particular disorder are not met. Instead, a maximum score (1 or 2) usually signifies that the individual meets the criteria for that disorder, with a score of 2 typically indicating a stronger or more definite endorsement of the disorder's symptoms, or a more severe presentation.
Symptom Check List (SCL-90) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  A measure of psychopathology symptoms and their intensity at a specific point in time. It includes 90 items that assess various symptom categories, such as anxiety, depression, and interpersonal sensitivity, among others. The overall score, known as the Global Severity Index (GSI), provides a measure of the overall psychological distress, and higher scores generally reflect greater symptom intensity and distress.
Toronto Alexithymia Scale (TAS - 20; Taylor & Bagby, 1992) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  It assesses difficulties in understanding, processing, or describing emotions. It consists of 20 items that assess emotional processing and expression. Global score ranges from 20 to 100, where 100 indicates the highest level of alexithymia.
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  A self-report scale measuring individual differences in the ability to identify, accept and manage emotional experiences. This measure help in understanding emotional dysregulation that might underlie the disorders. Global score ranges from 33 to 132, where 132 represents the highest level of difficulty in emotion regulation.
Multidimensional Perfectionism Scale (MPS; Hewitt & Flett, 2004) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  Measures the presence and extent of the perfectionism construct. It consists of 45 items, with each item rated on a scale from 1 to 7. A higher score indicates higher levels of perfectionism.
Perfectionistic Cognitions Inventory (PCI; Flett, Hewitt, Blankstein & Gray, 1998) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  Investigate the presence of perfectionist thoughts and cognitions. The Perfectionistic Cognitions Inventory consists of 15 items, each rated on a scale from 0 to 4. A higher score indicates greater concern with perfectionism.
Rosenberg Self-Exteem Scale (RSES; Rosenberg, 1965) | Time Frame: Change from baseline until after 20 sessions (approximately after 5 months), at the end of the treatment (approximately after 10 months) and in the following 3 months after treatment (approximately after 13 months).
  Assesses the subject's level of self-esteem. The global score ranges from 0 to 30, where higher scores indicate higher self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Dimaggio, Study Chair — Centro di Terapia Metacognitiva Interpersonale, Roma
Locations (2):
- Italy (2):
  - Centro Trattamento Integrato Disturbi Alimentari e Obesità, Verona, Italia
  - Centro Trattamento Integrato Disturbi Alimentari e Obesità, Verona, Verona

IPD SHARING:
Plan to Share IPD: Yes
Outcomes, age, gender
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 10 years
Access Criteria: Someone who has a request

REFERENCES:
- [Background] Accurso EC, Fitzsimmons-Craft EE, Ciao A, Cao L, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ, Wonderlich SA, Peterson CB. Therapeutic alliance in a randomized clinical trial for bulimia nervosa. J Consult Clin Psychol. 2015 Jun;83(3):637-42. doi: 10.1037/ccp0000021. Epub 2015 Apr 20. PMID 25894667
- [Background] Zipfel S, Wild B, Gross G, Friederich HC, Teufel M, Schellberg D, Giel KE, de Zwaan M, Dinkel A, Herpertz S, Burgmer M, Lowe B, Tagay S, von Wietersheim J, Zeeck A, Schade-Brittinger C, Schauenburg H, Herzog W; ANTOP study group. Focal psychodynamic therapy, cognitive behaviour therapy, and optimised treatment as usual in outpatients with anorexia nervosa (ANTOP study): randomised controlled trial. Lancet. 2014 Jan 11;383(9912):127-37. doi: 10.1016/S0140-6736(13)61746-8. Epub 2013 Oct 14. PMID 24131861
- [Background] Wilson GT, Fairburn CC, Agras WS, Walsh BT, Kraemer H. Cognitive-behavioral therapy for bulimia nervosa: time course and mechanisms of change. J Consult Clin Psychol. 2002 Apr;70(2):267-74. PMID 11952185
- [Background] Westwood H, Kerr-Gaffney J, Stahl D, Tchanturia K. Alexithymia in eating disorders: Systematic review and meta-analyses of studies using the Toronto Alexithymia Scale. J Psychosom Res. 2017 Aug;99:66-81. doi: 10.1016/j.jpsychores.2017.06.007. Epub 2017 Jun 11. PMID 28712432
- [Background] Watson HJ, Fursland A, Byrne S. Treatment engagement in eating disorders: who exits before treatment? Int J Eat Disord. 2013 Sep;46(6):553-9. doi: 10.1002/eat.22085. Epub 2013 Feb 25. PMID 23436476
- [Background] Treasure J, Cardi V, Leppanen J, Turton R. New treatment approaches for severe and enduring eating disorders. Physiol Behav. 2015 Dec 1;152(Pt B):456-65. doi: 10.1016/j.physbeh.2015.06.007. Epub 2015 Jun 6. PMID 26057573
- [Background] Treasure J, Sepulveda AR, MacDonald P, Whitaker W, Lopez C, Zabala M, Kyriacou O, Todd G. The assessment of the family of people with eating disorders. Eur Eat Disord Rev. 2008 Jul;16(4):247-55. doi: 10.1002/erv.859. PMID 18240125
- [Background] Thompson-Brenner H, Shingleton RM, Thompson DR, Satir DA, Richards LK, Pratt EM, Barlow DH. Focused vs. Broad enhanced cognitive behavioral therapy for bulimia nervosa with comorbid borderline personality: A randomized controlled trial. Int J Eat Disord. 2016 Jan;49(1):36-49. doi: 10.1002/eat.22468. Epub 2015 Dec 9. PMID 26649812
- [Background] Tatham M. The role of imagery-based techniques in cognitive-behavioural therapy for adults with eating disorders. Clin Psychol Rev. 2011 Nov;31(7):1101-9. doi: 10.1016/j.cpr.2011.06.008. Epub 2011 Jul 19. PMID 21820388
- [Background] Sodersten P, Bergh C, Leon M, Brodin U, Zandian M. Cognitive behavior therapy for eating disorders versus normalization of eating behavior. Physiol Behav. 2017 May 15;174:178-190. doi: 10.1016/j.physbeh.2017.03.016. Epub 2017 Mar 16. PMID 28322911
- [Background] Simpson S, Azam F, Brown S, Hronis A, Brockman R. The impact of personality disorders and personality traits on psychotherapy treatment outcome of eating disorders: A systematic review. Personal Ment Health. 2022 Aug;16(3):217-234. doi: 10.1002/pmh.1533. Epub 2021 Dec 5. PMID 34866357
- [Background] Simonsen S, Popolo R, Juul S, Frandsen FW, Sorensen P, Dimaggio G. Treating Avoidant Personality Disorder With Combined Individual Metacognitive Interpersonal Therapy and Group Mentalization-Based Treatment: A Pilot Study. J Nerv Ment Dis. 2022 Mar 1;210(3):163-171. doi: 10.1097/NMD.0000000000001432. PMID 34710894
- [Background] Semerari A, Colle L, Pellecchia G, Buccione I, Carcione A, Dimaggio G, Nicolo G, Procacci M, Pedone R. Metacognitive dysfunctions in personality disorders: correlations with disorder severity and personality styles. J Pers Disord. 2014 Dec;28(6):751-66. doi: 10.1521/pedi_2014_28_137. PMID 24689762
- [Background] Sassaroli S, Ruggiero GM. The role of stress in the association between low self-esteem, perfectionism, and worry, and eating disorders. Int J Eat Disord. 2005 Mar;37(2):135-41. doi: 10.1002/eat.20079. PMID 15732079
- [Background] Ruggiero GM, Levi D, Ciuna A, Sassaroli S. Stress situation reveals an association between perfectionism and drive for thinness. Int J Eat Disord. 2003 Sep;34(2):220-6. doi: 10.1002/eat.10191. PMID 12898558
- [Background] Rania M, Monell E, Sjolander A, Bulik CM. Emotion dysregulation and suicidality in eating disorders. Int J Eat Disord. 2021 Mar;54(3):313-325. doi: 10.1002/eat.23410. Epub 2020 Nov 18. PMID 33205495
- [Background] Poulsen S, Lunn S, Daniel SI, Folke S, Mathiesen BB, Katznelson H, Fairburn CG. A randomized controlled trial of psychoanalytic psychotherapy or cognitive-behavioral therapy for bulimia nervosa. Am J Psychiatry. 2014 Jan;171(1):109-16. doi: 10.1176/appi.ajp.2013.12121511. PMID 24275909
- [Background] Popolo R, MacBeth A, Lazzerini L, Brunello S, Venturelli G, Rebecchi D, Morales MF, Dimaggio G. Metacognitive interpersonal therapy in group versus TAU + waiting list for young adults with personality disorders: Randomized clinical trial. Personal Disord. 2022 Nov;13(6):619-628. doi: 10.1037/per0000497. Epub 2021 Aug 12. PMID 34383540
- [Background] Popolo R, MacBeth A, Brunello S, Canfora F, Ozdemir E, Rebecchi D, Toselli C, Venturelli G, Salvatore G, Dimaggio G. Metacognitive interpersonal therapy in group: a feasibility study. Res Psychother. 2018 Dec 18;21(3):338. doi: 10.4081/ripppo.2018.338. eCollection 2018 Dec 19. PMID 32913773
- [Background] Misso D, Velotti P, Pasetto A, Dimaggio G. Treating intimate partner violence with metacognitive interpersonal therapy: The case of Aaron. J Clin Psychol. 2022 Jan;78(1):50-66. doi: 10.1002/jclp.23294. Epub 2021 Dec 20. PMID 34927730
- [Background] Neumark-Sztainer D, Hannan PJ. Weight-related behaviors among adolescent girls and boys: results from a national survey. Arch Pediatr Adolesc Med. 2000 Jun;154(6):569-77. doi: 10.1001/archpedi.154.6.569. PMID 10850503
- [Background] Murphy R, Straebler S, Cooper Z, Fairburn CG. Cognitive behavioral therapy for eating disorders. Psychiatr Clin North Am. 2010 Sep;33(3):611-27. doi: 10.1016/j.psc.2010.04.004. PMID 20599136
- [Background] Meneguzzo P, Cazzola C, Castegnaro R, Buscaglia F, Bucci E, Pillan A, Garolla A, Bonello E, Todisco P. Associations Between Trauma, Early Maladaptive Schemas, Personality Traits, and Clinical Severity in Eating Disorder Patients: A Clinical Presentation and Mediation Analysis. Front Psychol. 2021 Mar 31;12:661924. doi: 10.3389/fpsyg.2021.661924. eCollection 2021. PMID 33868136
- [Background] McIntosh VV, Carter FA, Bulik CM, Frampton CM, Joyce PR. Five-year outcome of cognitive behavioral therapy and exposure with response prevention for bulimia nervosa. Psychol Med. 2011 May;41(5):1061-71. doi: 10.1017/S0033291710001583. PMID 20810005
- [Background] Martinussen M, Friborg O, Schmierer P, Kaiser S, Overgard KT, Neunhoeffer AL, Martinsen EW, Rosenvinge JH. The comorbidity of personality disorders in eating disorders: a meta-analysis. Eat Weight Disord. 2017 Jun;22(2):201-209. doi: 10.1007/s40519-016-0345-x. Epub 2016 Dec 19. PMID 27995489
- [Background] Maher A, Cason L, Huckstepp T, Stallman H, Kannis-Dymand L, Millear P, Mason J, Wood A, Allen A. Early maladaptive schemas in eating disorders: A systematic review. Eur Eat Disord Rev. 2022 Jan;30(1):3-22. doi: 10.1002/erv.2866. Epub 2021 Oct 12. PMID 34636456
- [Background] Le Grange D, Eckhardt S, Dalle Grave R, Crosby RD, Peterson CB, Keery H, Lesser J, Martell C. Enhanced cognitive-behavior therapy and family-based treatment for adolescents with an eating disorder: a non-randomized effectiveness trial. Psychol Med. 2020 Dec 3;52(13):1-11. doi: 10.1017/S0033291720004407. Online ahead of print. PMID 33267919
- [Background] Inchausti F, Garcia-Poveda NV, Ballesteros-Prados A, Ortuno-Sierra J, Sanchez-Reales S, Prado-Abril J, Aldaz-Armendariz JA, Mole J, Dimaggio G, Ottavi P, Fonseca-Pedrero E. The Effects of Metacognition-Oriented Social Skills Training on Psychosocial Outcome in Schizophrenia-Spectrum Disorders: A Randomized Controlled Trial. Schizophr Bull. 2018 Oct 17;44(6):1235-1244. doi: 10.1093/schbul/sbx168. PMID 29267940
- [Background] Harris BA, Scharff A, Smith M, Brooks G, Thompson-Brenner H, Boswell JF. Trajectories of interpersonal problems in residential eating disorder treatment: Exploring the influence of primary diagnosis. Clin Psychol Psychother. 2023 Mar;30(2):302-316. doi: 10.1002/cpp.2795. Epub 2022 Nov 9. PMID 36303012
- [Background] Griffen TC, Naumann E, Hildebrandt T. Mirror exposure therapy for body image disturbances and eating disorders: A review. Clin Psychol Rev. 2018 Nov;65:163-174. doi: 10.1016/j.cpr.2018.08.006. Epub 2018 Aug 29. PMID 30223161
- [Background] Grenon R, Carlucci S, Brugnera A, Schwartze D, Hammond N, Ivanova I, Mcquaid N, Proulx G, Tasca GA. Psychotherapy for eating disorders: A meta-analysis of direct comparisons. Psychother Res. 2019 Oct;29(7):833-845. doi: 10.1080/10503307.2018.1489162. Epub 2018 Jun 29. PMID 29958509
- [Background] Geller J, Srikameswaran S, Cockell SJ, Zaitsoff SL. Assessment of shape- and weight-based self-esteem in adolescents. Int J Eat Disord. 2000 Nov;28(3):339-45. doi: 10.1002/1098-108x(200011)28:33.0.co;2-r. PMID 10942921
- [Background] Garner DM, Garfinkel PE. The Eating Attitudes Test: an index of the symptoms of anorexia nervosa. Psychol Med. 1979 May;9(2):273-9. doi: 10.1017/s0033291700030762. PMID 472072
- [Background] Frostad S, Danielsen YS, Rekkedal GA, Jevne C, Dalle Grave R, Ro O, Kessler U. Implementation of enhanced cognitive behaviour therapy (CBT-E) for adults with anorexia nervosa in an outpatient eating-disorder unit at a public hospital. J Eat Disord. 2018 May 29;6:12. doi: 10.1186/s40337-018-0198-y. eCollection 2018. PMID 29854400
- [Background] Frostad S, Calugi S, Engen CBN, Dalle Grave R. Enhanced cognitive behaviour therapy (CBT-E) for severe and extreme anorexia nervosa in an outpatient eating disorder unit at a public hospital: a quality-assessment study. J Eat Disord. 2021 Nov 2;9(1):143. doi: 10.1186/s40337-021-00499-1. PMID 34727976
- [Background] Fairburn CG, Patel V. The global dissemination of psychological treatments: a road map for research and practice. Am J Psychiatry. 2014 May;171(5):495-8. doi: 10.1176/appi.ajp.2013.13111546. No abstract available. PMID 24788281
- [Background] Fairburn CG, Doll HA, Welch SL, Hay PJ, Davies BA, O'Connor ME. Risk factors for binge eating disorder: a community-based, case-control study. Arch Gen Psychiatry. 1998 May;55(5):425-32. doi: 10.1001/archpsyc.55.5.425. PMID 9596045
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Eielsen HP, Vrabel K, Hoffart A, Ro O, Rosenvinge JH. Reciprocal relationships between personality disorders and eating disorders in a prospective 17-year follow-up study. Int J Eat Disord. 2022 Dec;55(12):1753-1764. doi: 10.1002/eat.23823. Epub 2022 Oct 10. PMID 36214278
- [Background] Dalle Grave R, Calugi S, Conti M, Doll H, Fairburn CG. Inpatient cognitive behaviour therapy for anorexia nervosa: a randomized controlled trial. Psychother Psychosom. 2013;82(6):390-8. doi: 10.1159/000350058. Epub 2013 Sep 20. PMID 24060628
- [Background] Dalle Grave R, Calugi S, Doll HA, Fairburn CG. Enhanced cognitive behaviour therapy for adolescents with anorexia nervosa: an alternative to family therapy? Behav Res Ther. 2013 Jan;51(1):R9-R12. doi: 10.1016/j.brat.2012.09.008. Epub 2012 Oct 4. PMID 23123081
- [Background] Dahlenburg SC, Gleaves DH, Hutchinson AD. Anorexia nervosa and perfectionism: A meta-analysis. Int J Eat Disord. 2019 Mar;52(3):219-229. doi: 10.1002/eat.23009. Epub 2019 Jan 11. PMID 30632629
- [Background] Cruz-Saez S, Pascual A, Wlodarczyk A, Echeburua E. The effect of body dissatisfaction on disordered eating: The mediating role of self-esteem and negative affect in male and female adolescents. J Health Psychol. 2020 Jul;25(8):1098-1108. doi: 10.1177/1359105317748734. Epub 2018 Aug 11. PMID 30101609
- [Background] Costa S, Hausenblas HA, Oliva P, Cuzzocrea F, Larcan R. Maladaptive perfectionism as mediator among psychological control, eating disorders, and exercise dependence symptoms in habitual exerciser. J Behav Addict. 2016 Mar;5(1):77-89. doi: 10.1556/2006.5.2016.004. PMID 28092194
- [Background] Cooper Z, Fairburn CG. The Evolution of "Enhanced" Cognitive Behavior Therapy for Eating Disorders: Learning From Treatment Nonresponse. Cogn Behav Pract. 2011 Aug;18(3):394-402. doi: 10.1016/j.cbpra.2010.07.007. PMID 23814455
- [Background] Cheli S, Cavalletti V, Flett GL, Hewitt PL. Perfectionism unbound: An integrated individual and group intervention for those hiding imperfections. J Clin Psychol. 2022 Aug;78(8):1624-1636. doi: 10.1002/jclp.23365. Epub 2022 Apr 29. PMID 35486835
- [Background] Carlson L, Steward T, Aguera Z, Mestre-Bach G, Magana P, Granero R, Jimenez-Murcia S, Claes L, Gearhardt AN, Menchon JM, Fernandez-Aranda F. Associations of food addiction and nonsuicidal self-injury among women with an eating disorder: A common strategy for regulating emotions? Eur Eat Disord Rev. 2018 Nov;26(6):629-637. doi: 10.1002/erv.2646. Epub 2018 Oct 15. PMID 30318670
- [Background] Button EJ, Sonuga-Barke EJ, Davies J, Thompson M. A prospective study of self-esteem in the prediction of eating problems in adolescent schoolgirls: questionnaire findings. Br J Clin Psychol. 1996 May;35(2):193-203. doi: 10.1111/j.2044-8260.1996.tb01176.x. PMID 8773797
- [Background] Butler RM, Heimberg RG. Exposure therapy for eating disorders: A systematic review. Clin Psychol Rev. 2020 Jun;78:101851. doi: 10.1016/j.cpr.2020.101851. Epub 2020 Mar 21. PMID 32224363
- [Background] Brugnera A, Lo Coco G, Salerno L, Sutton R, Gullo S, Compare A, Tasca GA. Patients with Binge Eating Disorder and Obesity have qualitatively different interpersonal characteristics: Results from an Interpersonal Circumplex study. Compr Psychiatry. 2018 Aug;85:36-41. doi: 10.1016/j.comppsych.2018.06.008. Epub 2018 Jun 21. PMID 29960139
- [Background] Boone L, Braet C, Vandereycken W, Claes L. Are maladaptive schema domains and perfectionism related to body image concerns in eating disorder patients? Eur Eat Disord Rev. 2013 Jan;21(1):45-51. doi: 10.1002/erv.2175. Epub 2012 May 3. PMID 22556040
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Basile B, Novello C, Calugi S, Dalle Grave R, Mancini F. Childhood Memories in Eating Disorders: An Explorative Study Using Diagnostic Imagery. Front Psychol. 2021 Jul 22;12:685194. doi: 10.3389/fpsyg.2021.685194. eCollection 2021. PMID 34367006
- [Background] Atwood ME, Friedman A. A systematic review of enhanced cognitive behavioral therapy (CBT-E) for eating disorders. Int J Eat Disord. 2020 Mar;53(3):311-330. doi: 10.1002/eat.23206. Epub 2019 Dec 16. PMID 31840285
- [Background] Arcelus J, Haslam M, Farrow C, Meyer C. The role of interpersonal functioning in the maintenance of eating psychopathology: a systematic review and testable model. Clin Psychol Rev. 2013 Feb;33(1):156-67. doi: 10.1016/j.cpr.2012.10.009. Epub 2012 Nov 10. PMID 23195616
- [Background] Anderson LK, Claudat K, Cusack A, Brown TA, Trim J, Rockwell R, Nakamura T, Gomez L, Kaye WH. Differences in emotion regulation difficulties among adults and adolescents across eating disorder diagnoses. J Clin Psychol. 2018 Oct;74(10):1867-1873. doi: 10.1002/jclp.22638. Epub 2018 May 13. PMID 29756232
- [Background] Anderson DA, Maloney KC. The efficacy of cognitive-behavioral therapy on the core symptoms of bulimia nervosa. Clin Psychol Rev. 2001 Oct;21(7):971-88. doi: 10.1016/s0272-7358(00)00076-3. PMID 11584518
- [Background] Aloi M, Rania M, Carbone EA, Caroleo M, Calabro G, Zaffino P, Nicolo G, Carcione A, Coco GL, Cosentino C, Segura-Garcia C. Metacognition and emotion regulation as treatment targets in binge eating disorder: a network analysis study. J Eat Disord. 2021 Feb 15;9(1):22. doi: 10.1186/s40337-021-00376-x. PMID 33588943
- [Background] Aloi M, Rania M, Caroleo M, Carbone EA, Fazia G, Calabro G, Segura-Garcia C. How are early maladaptive schemas and DSM-5 personality traits associated with the severity of binge eating? J Clin Psychol. 2020 Mar;76(3):539-548. doi: 10.1002/jclp.22900. Epub 2019 Nov 16. PMID 31733127
- [Background] Allen KL, Fursland A, Raykos B, Steele A, Watson H, Byrne SM. Motivation-focused treatment for eating disorders: a sequential trial of enhanced cognitive behaviour therapy with and without preceding motivation-focused therapy. Eur Eat Disord Rev. 2012 May;20(3):232-9. doi: 10.1002/erv.1131. Epub 2011 Jul 26. PMID 21793108
- [Background] Agras WS, Walsh T, Fairburn CG, Wilson GT, Kraemer HC. A multicenter comparison of cognitive-behavioral therapy and interpersonal psychotherapy for bulimia nervosa. Arch Gen Psychiatry. 2000 May;57(5):459-66. doi: 10.1001/archpsyc.57.5.459. PMID 10807486